

## **CLINICAL TRIAL PROTOCOL**

## **PROTOCOL TITLE:**

Eradicating minimal residual disease using "off the shelf" Natural Killer (NK) cells for advanced nasopharyngeal cancer

PROTOCOL NUMBER: 001

**CIRB NUMBER:** 2024-2264

NCT NUMBER: NCT07247201

**PROTOCOL VERSION:** Version 6

**PROTOCOL DATE**: 21 October 2025

## PRINCIPAL INVESTIGATOR:

Lim Chwee Ming

## SITE PRINCIPAL INVESTIGATOR:

Lim Chwee Ming, Senior Consultant, SGH

## **TABLE OF CONTENT**

| 1 BAC | CKGROUND AND RATIONALE | 6 |
|-------|-------------------------------------------------------|----|
| 1.1 | GENERAL INTRODUCTION | 6 |
| 1.2 | RATIONALE AND JUSTIFICATION FOR THE STUDY | 7 |
| 1.2.1 | RATIONALE FOR THE STUDY PURPOSE | 7 |
| 1.2.2 | RATIONALE FOR DOSES SELECTED | 8 |
| 1.2.3 | RATIONALE FOR STUDY POPULATION | 8 |
| 1.2.4 | RATIONALE FOR STUDY DESIGN | 8 |
| 2 HYF | POTHESIS AND OBJECTIVES | 9 |
| 2.1 | HYPOTHESIS | 9 |
| 2.2 | PRIMARY OBJECTIVES | 9 |
| 2.3 | SECONDARY OBJECTIVES | 9 |
| 2.4 | POTENTIAL RISKS AND BENEFITS: | 9 |
| 2.4.1 | POTENTIAL RISKS | 9 |
| 2.4.2 | POTENTIAL BENEFITS | 9 |
| 3 STU | IDY POPULATION | 9 |
| 3.1 | LIST THE NUMBER AND NATURE OF SUBJECTS TO BE ENROLLED | 9 |
| 3.2 | CRITERIA FOR RECRUITMENT AND RECRUITMENT PROCESS | 10 |
| 3.3 | INCLUSION CRITERIA | 10 |
| 3.4 | EXCLUSION CRITERIA | 10 |
| 3.5 | SUBJECT REPLACEMENT | 10 |
| 4 STU | IDY DESIGN | 10 |
| 4.1 | RANDOMISATION AND BLINDING | 12 |
| 4.2 | CONTRACEPTION AND PREGNANCY TESTING | 13 |
| 4.3 | STUDY VISITS AND PROCEDURES | 13 |
| 4.3.1 | SCREENING VISITS AND PROCEDURES | 15 |
| 4.3.2 | STUDY VISITS AND PROCEDURES | 15 |
| 4.3.3 | FINAL STUDY VISIT: | 18 |
| 4.3.4 | POST STUDY FOLLOW UP AND PROCEDURES | 18 |
| 4.4 | DISCONTINUATION/WITHDRAWAL | 18 |

| 4.4.1 | 1 DISCONTINUATION CRITERIA18 |
|---|---|
| 4.4.2 | 2 DISCONTINUATION VISIT AND PROCEDURES18 |
| 5 | TRIAL MATERIALS |
| 5.1 | TRIAL PRODUCT (S)19 |
| 5.1.1 | 1. CELL SOURCE |
| 5.1.2 | 2 SCREENING AND PRE-DONATION REQUIREMENTS19 |
| 5.1.3 | 3 INFECTIOUS DISEASE TESTING19 |
| 5.1.4 | 4. COLLECTION AND HANDLING19 |
| 5.1.5 | 5. ALLOGENEIC NK CELLS |
| 5.2 | STORAGE AND PRODUCT ACCOUNTABILITY24 |
| 6 | TREATMENT25 |
| 6.1 | RATIONALE FOR SELECTION OF DOSE25 |
| 6.2 | STUDY DRUG FORMULATIONS26 |
| 6.3 | STUDY DRUG ADMINISTRATION26 |
| 6.4 | SPECIFIC RESTRICTIONS / REQUIREMENTS26 |
| 6.5 | MONITORING REQUIREMENTS26 |
| 7.1 🛭 | DEFINITIONS27 |
| 7.2<br>(SAE | COLLECTING, RECORDING AND REPORTING OF SERIOUS ADVERSE EVENTS ES) TO CIRB |
| 7.3<br>(SAE | COLLECTING, RECORDING AND REPORTING OF SERIOUS ADVERSE EVENTS ES) TO THE HEALTH SCIENCES AUTHORITY (HSA)28 |
| 7.4<br>(ALL | KNOWN OR POTENTIAL ADVERSE EVENT RELATED TO POST-INFUSION OF IP LONK1) |
| 7.5<br>INFU | KNOWN OR POTENTIAL SERIOUS ADVERSE EVENT RELATED TO POST-<br>USION OF IP (ALLONK1)30 |
| 7.6 | MANAGEMENT OF AE AND SAE31 |
| 7.7 | SAFETY MONITORING PLAN32 |
| 7.8 | COMPLAINT HANDLING32 |
| 8 | DATA ANALYSIS |
| 8.1 | DATA QUALITY ASSURANCE32 |
| 8.2 | DATA ENTRY AND STORAGE32 |
| 9 | SAMPLE SIZE AND STATISTICAL METHODS32 |

| 9.1 | DETERMINATION OF SAMPLE SIZE | 32 |
|--------|---------------------------------------------|----|
| 9.2 | STATISTICAL AND ANALYTICAL PLANS | 33 |
| 9.3 | INTERIM ANALYSES | 38 |
| 10 D | IRECT ACCESS TO SOURCE DATA/DOCUMENTS | 38 |
| 11 Q | UALITY CONTROL AND QUALITY ASSURANCE | 38 |
| 12 E | THICAL CONSIDERATIONS | 38 |
| 12.1 | INFORMED CONSENT | 39 |
| 12.2 | CONFIDENTIALITY OF DATA AND PATIENT RECORDS | 39 |
| 13 PI | UBLICATIONS | 39 |
| 14 R | ETENTION OF TRIAL DOCUMENTS | 39 |
| 15 F | UNDING AND INSURANCE | 39 |
| LIST O | F ATTACHMENTS | 40 |
| APPE | NDIX 1 STUDY SCHEDULE | 40 |
| REFE | RENCES | 43 |

#### PROTOCOL SIGNATURE PAGE

Protocol Title: Eradicating minimal residual disease using "off the shelf" Natural Killer (NK) cells

for advanced nasopharyngeal cancer

**Protocol Number: 001** 

Protocol Version/ Date: Version 6 / 21 October 2025

Sponsor Name: National Medical Research Council under the CSA-INV grant

**Study Site(s):** Singapore General Hospital (SGH)

## **Declaration of Investigator**

I confirm that I have read the above-mentioned protocol and its attachments. I agree to conduct the described trial in compliance with all stipulations of the protocol, regulations and ICH E6 Guideline for Good Clinical Practice (GCP).

Principal Investigator: Lim Chwee Ming

Title: Senior Consultant, SGH

Principal Investigator Signature:

Date: 31 October 2025

Site Principal Investigator: Lim Chwee Ming

Title: Senior Consultant, SGH

Site Principal Investigator

Signature:

Date: 31 October 2025

#### 1 BACKGROUND AND RATIONALE

Nasopharyngeal carcinoma (NPC) is an aggressive head and neck cancer, primarily endemic in Singapore, Southeast Asia, Southern China and North Africa. A large majority (~70%) of NPC patients present with locally advanced disease at diagnosis and carry a high risk of recurrence (~30%) following definitive chemoradiotherapy (CRT). These relapses are highly lethal and current chemotherapies can prolong progressive-free survival by 6-8 months only. To reduce NPC-related mortality, preventive strategies aiming to reduce the risk of relapses with treatment intensification upfront should be more effective than delivering treatments after relapses have occurred.

Intensifying treatment in locally advanced NPC patients using adjuvant chemotherapy following conventional CRT is often not well-tolerated, given that these patients are still recuperating from the acute CRT toxicities. Conversely, immunotherapy options, such as cell-based therapy and immune checkpoint inhibitor, are good candidates of adjuvant treatments because they are very well-tolerated even when combined with chemotherapy. In line with this notion, our preliminary results have shown that the addition of functional NK cells to standard chemotherapy improved the prognostic outcome from chemotherapy alone based on the decrease in tumor growth rate and the final tumor volume. Therefore, this clinical trial is to validate if addition of NK infusion to NPC standard of care can reduce relapses and metastasis. Since NPC is ubiquitously associated with the Epstein Barr Virus (EBV) infection, detectable post-treatment circulating EBV-DNA is well-documented to represent minimal residue disease (MRD), which portends a worse prognosis. Therefore, complete eradication of remaining circulating EBV-DNA NPC cells would eliminate MRD following treatment, thereby reducing the risk of future relapses.

With these rationale in mind, our aim is to perform a dose escalating clinical trial to identify the maximum tolerate dose of allogeneic "off the shelf" NK cells integrated into the current standard of care treatment of advanced NPC patients; and investigate if addition of allogeneic "off the shelf" NK cells in the concurrent and adjuvant setting can reduce the probability of having detectable plasma EBV-DNA after definitive treatment.

#### 1.1 General Introduction

NK cells is a member of the innate lymphoid cells (ILC) that is able to recognize and eradicate tumor cells without engaging MHC class I [1, 2]. A critical component of our innate immune system, NK cells is our first line of defence against carcinogenesis by their constant surveillance and elimination of circulating tumor cells [3, 4]. For the past decade, NK cells are constantly being explored as a new cell therapy in cancer treatment [5, 6]. The success in using NK cells to eliminate leukaemia has render much promise and merits to extend its use to treat solid tumor. In the past five years, several Phase I studies were being reported demonstrating good tolerance to the dosage of 0.5 to 3 billion allogeneic NK cells (derived from in-vitro expansion from PBMC) in cancer patients with no significant GVHD symptoms [7-10]. In addition, a study two years ago documenting the success in eliminating brain metastasis from NPC after failed chemotherapy using periodic infusion of 2 billion of allogeneic NK cells [11].

## 1.2 Rationale and Justification for the Study

This is a phase 1 leading to a Phase 2 clinical trial investigating addition of allogeneic NK cells to conventional CRT for locally advanced NPC patients. We hypothese <u>that allogeneic NK cells are</u> well-tolerated and safe when used in combination with conventional CRT in treating locally advanced NPC and lead to elimination of post-treatment circulating EBV-DNA from the current 25-30% to 10% among locally advanced NPC patients.

From a mechanistic perspective, during concurrent CRT, the NPC tumor will be killed and fragments of the EBV positive NPC tumor cells will be released into the circulation. In usual instance, the host circulating NK cells will be responsible to "mop" up these circulating NPC cells that may be still viable. However, due to the effects of immune suppression from chemotherapy, some of these circulating NPC cells may not be adequately eliminated, resulting in missed opportunity to completely eradicate these circulating NPC cells. These viable cells may enter into dormancy and only to re-emerge subsequently as clinically evident cancer relapses. Therefore, in our trial design, we have purposefully integrate the use of allogeneic NK cells during the concurrent (2 doses) and adjuvant (4 doses) phase. We hypothese that by supplementing NK cells in these critical phases, the circulating NPC cells can be effectively killed and completely eliminated. Additionally, we also have highly sensitive plasma EBV-DNA assays that will allow us to measure and track the circulating NPC cells during this trial. A summary of our mechanistic explanation of our study is presented in Figure 1.



Figure 1:

Mechanistic explanation to leverage on allogeneic NK cells to mop up circulating EBV-NPC cells following concurrent chemoradiotherapy. The lysed NPC cells following NK cell mediated cytotoxicity can further promote anti-NPC T cell responses from NK cell-dendritic cell cross presentation

## 1.2.1 Rationale for the Study Purpose

A large majority (~70%) of Nasopharyngeal Carcinoma (NPC) patients present with <u>locally advanced disease</u> at diagnosis <u>carry a high risk of recurrence (~30%)</u> following definitive chemoradiotherapy (CRT). Preventive strategies with treatment intensification upfront should be more effective than delivering treatments after relapses have occurred. However, Intensifying conventional CRT as adjuvant treatment in locally advanced NPC patients is often not well-tolerated, given that these patients are still recuperating from acute CRT toxicities. Conversely, NK cell therapy has shown to be very well-tolerated when use as sole therapeutic in cancer patients. Together with their capacity to eliminate tumor cells without engaging MHC class I or prior antigenic engagement, allogeneic NK cell is expected to be an ideal adjuvant immunotherapy to be combined with chemotherapy. To date however, such combinatory therapeutic approach towards cancer treatment has not been investigated for NPC. In this clinical trial, we proposed a phase I study to

determine the maximum Tolerated Dose (MTD) of allogeneic NK cells to be used in the trial, leading to a phase 2 study to evaluate the efficacy of such combined treatment approach on reducing cancer recurrence for NPC patients.

#### 1.2.2 Rationale for Doses Selected

We anticipate the maximum Tolerated Dose (MTD) to be between  $0.8 \times 10^7$  to  $1.8 \times 10^7$  NK cells/kg (equivalent to approximately 0.5 to 1.0 billion NK cells) because this dosage range of allogeneic NK cells has been shown to be safe and feasible among several Phase I clinical trials [7-10]. Therefore, our team has adopted in this Phase I trial the same dosing regime in a carefully escalated manner.

## 1.2.3 Rationale for Study Population

We are selecting only locally advanced NPC patients who are at high risk of developing relapses in the future. Based on previous studies across many tertiary centers, locally advanced NPC patients (ie Stage III-IVA/B, T1-4, N1-3, M0) are at higer risk of future cancer relapse following current standard of care treatment with concurrent CRT. With a larger tumor burden, we believe that addition of allogeneic NK cells can help to "mop" up the circulating EBV NPC cells during and after the standard of care CRT treatment.

## 1.2.4 Rationale for Study Design

In Phase 1 study, we will determine the MTD using the Bayesian Model Averaging continual reassessment method (BMA-CRM) study design [12, 13] where <u>5 doses (0.5x10<sup>7</sup>, 0.8x10<sup>7</sup>, 1.1x10<sup>7</sup>, 1.4x10<sup>7</sup> and 1.8x 10<sup>7</sup> cells/Kg) of NK cells will be evaluated. The primary goal of the BMA-CRM is to identify the maximum tolerated dose (MTD) of NK cells to be infused. An anticipated size of 6 patients will be accrued for the Phase 1 study. If the MTD is achieved earlier with smaller cohort of patients, we will proceed with phase 2 portion without having to complete the projected 25 patients accrual on the phase 1 design.</u>

The Phase 2 study is a single-arm trial derived from the anticipated proportion of locally advanced NPC patients (25-30%) who will continue to present with detectable circulating EBV-DNA following standard of care CRT paradigm. We hypothesize that in this single arm trial, adding allogeneic NK cells will completely eliminate the proportion of patients with detectable circulating EBV-DNA from 25-30% to 10%.

Hence, applying the one proportion Z-score test, a sample size of 9 will achieve 80.5% power to detect a difference (P1-P0) of -0.2500% using a one-sided exact test with a significance level (alpha) of 0.05. Assume the withdrawal rate at 0.2 (20%), the total sample size is estimated at 12.

In our phase 1 design, at least 6 patients will be treated at our MTD of allogenic NK cells, meaning that additional 25 patients will be accrued in the phase 2 trial.

#### 2 HYPOTHESIS AND OBJECTIVES

## 2.1 Hypothesis

The hypothesis of this trial is allogeneic NK cells wil be well-tolerated and safe when used in combination with conventional CRT in locally advanced NPC patients leading to the elimination of post-treatment circulating EBV-DNA from the current 30% to 10% in locally advanced NPC patients.

## 2.2 Primary Objectives

The primary objective of this trial is to determine the MTD of allogeneic NK cells when used with concurrent CRT in advanced NPC patients.

## 2.3 Secondary Objectives

The secondary objective of this trial is to determine if adding allogeneic NK cells to NPC standard of care CRT treatment paradigm can decrease the percentage of NPC patients' conversion to undetectable plasma EBV-DNA levels from 30 to 10%. The time to relapse will also be measured as an additional secondary endpoint.

#### 2.4 Potential Risks and Benefits:

#### 2.4.1 Potential Risks

Allogeneic NK cells are generally safe to administer with minimal toxicities reported. The risk of graft versus host disease (GVHD) are generally very low, in comparison with T cell therapy. As part of the release criteria of our NK cells, we will ensure that the minimum purity of NK cells to be at least 90%, before these cells are administered to patients. Once our MTD of NK cells is ascertained, this dose will be delivered in the phase 2 portion of the study.

#### 2.4.2 Potential Benefits

Integrating NK cells into CRT can potentially reduce the risk of future cancer relapse of NPC patients receiving definitive treatment. This risk can be objectively measured using circulating plasma EBV-DNA post treatment. Therefore, in this trial, we will measure the circulating plasma EBV-DNA longitudinally and ascertain if the addition of NK cells can reduce the risk of having detectable plasma EBV-DNA following current standard of care treatment of CRT.

#### 3 STUDY POPULATION

## 3.1 List The Number and Nature of Subjects to be Enrolled

We intend to accrue 31 patients for this Phase I leading to Phase II study.

These patients are newly diagnosed advanced non-metastatic NPC patients who are at high risk of future cancer relapse.

## 3.2 Criteria for Recruitment and Recruitment Process

We plan to enrol up to 31 patients (6 in phase 1, 25 in phase 2) within a period of 24-36 months, from Singapore General Hospital, Sengkang General Hospital, Changi General Hospital and National Cancer Center (NCC) Singapore.

Newly diagnosed NPC patients with Stage III-IVA/B (T1-4, N1-3, M0)) disease and planned to start standard of care treatment will be identified and recruited. The specific inclusion and exclusion criteria are summarized in section 3.3 and 3.4 respectively. Patients satisfying the inclusion criteria will be approached for consent to participate in this clinical trial.

#### 3.3 Inclusion Criteria

- Age 21-80
- NPC Stage III-IVA/B (T1-4, N1-3, M0)
- Able to tolerate conventional CRT
- Detectable EBV level at diagnosis
- Adequate organ function
  - ANC ≥ 1500/µL
  - o Platelet count ≥ 100,000/µL
  - o Creatinine clearance ≥60ml/minute
  - o Total bilirubin ≤ 1.5 x upper limit normal (ULN)
  - o AST ≤ 2 x upper limit normal
  - o ALT ≤ 2 x upper limit normal
- ECOG performance status of 0-1

#### 3.4 Exclusion Criteria

- Presence of Autoimmune Disease
- Any conditions resulting in Immunocompromised state (Drug induced)
- ECOG performance status ≥ 2
- Poor organ function
- Lactating or pregnant
- Serious concomitant disorders that would compromise the safety of the patient or compromise the patients ability to complete the study.

#### 3.5 Subject Replacement

An accrued patient who fails to receive the first NK cell infusion during treatment will be considered non-evaluable, and will be replaced.

#### 4 STUDY DESIGN

This Clinical Trial comprised of a Phase 1 study leading to a single arm Phase 2 study.

<u>For the Phase 1 study:</u> Determination of the maximum tolerated dose (MTD) using Continual Reassessment Method (CRM).

1. Doses to be evaluated  $(0.5x10^7, 0.8x10^7, 1.1x10^7, 1.4x10^7)$  and  $1.8x 10^7$  cells/kg).

- 2. The starting dose to be evaluated is 0.8x10<sup>7</sup> cells/kg.
- 3. Dose Limiting Toxicity (DLT): Grade 3 to 5 toxicities (using Common Terminology Criteria for Adverse Events CTCAE).
- 4. Target Toxicity Limit (TTL): maximum probability of DLT occurring before rejecting the dose is set at 30% (0.3).



For every case of DLT encountered, the toxicity limit will be reassessed to ascertain whether it has reached the TTL. In the instance when the cohort size is reached and the toxicity limit < or = TTL, the dose will be escalated for MTD evaluation. Otherwise, if the toxicity limit > TTL, current dose will be rejected as MTD and the dose will be de-escalated for MTD evaluation. When the toxicity limit is very low, the dose escalation for MTD evaluated can be accelerated. i.e. escalating from dose 2 to 4 as shown in Figure 2. When 6 patients treated at our set MTD do not develop grade 3-5 toxicities, the phase 1 portion of our study will be deemed to be completed, and then the set MTD will be accepted. Every accrued patients involved in MTD evaluation will undergo the standard NPC treatment with the NK cells infusion dose set at the previously evaluated dose.

#### For the Phase 2 study:

- 5. Standard Chemoradiotherapy will be implemented to every accrued NPC patients.
- 6. The dose of NK cells used will be set at MTD or the dose where the patient is subjected during Phase 1.
- 7. NK cells infusion will be carried out 1 time/week at week 3, 6, 7, 8, 9 and 10.
- 8. Interlukin-2 (200U/ml) will be delivered together with the NK cells in Plasma-Lyte 148 supplemented with 2% Human Serum Albumin (HSA).
- 9. Primary endpoint is set at the percentage of patients with detectable post-treatment circulating EBV-DNA has decreased from 30% to 10%.

10. Secondary endpoint is in determining the change in patient survival and recurrence rate within 24-36 months post-treatment under this new treatment regimen when compare with historic cohorts under standard treatments.



The treatment regimen for the single arm Phase 2 study is showed in Figure 3. The 6 doses of NK cells will be infused once a week at specific week of treatment into every accrued patient. IL-2 will be combined with NK cells in Plasma-Lyte148 supplementd with 2% HSA and infused concurrently as a single product in one infusion bag . The NK cells are derived from healthy donors PBMC. At week 9, patients whose circulating EBV-DNA have decreased but not to undetectable level have the option of undergoing an additional 4 doses of NK cells infusion at week 12 to 15.

## 4.1 Randomisation and Blinding

This Phase 1 leading to Phase 2 trial is a single arm clinical trial. There will not be any randomization or blinding requFired.

## 4.2 Contraception and Pregnancy Testing

For this trial, pregnant woman is a criterion for exclusion. Pregnant patients are excluded from receiving chemoradiotherapy as the standard of care CRT treatment. All females of reproductive age will be undergoing a pregnancy test as standard clinical care prior to receive CRT.

## 4.3 Study Visits and Procedures

A table of scheduled study assessments for screening is provided in Table 1, Table 2 and Appendix 1. The Study will conclude ~ 4 months after accrual. Patients following treatment will be followed up as per normal standard of care by their treating physician at both National Cancer Center (NCC) and their respective treating ENT specialists. All assessments must be performed and documented in the medical record for each patient.

Screening evaluations will be performed  $\leq$  28 days before enrollment. Patients who agree to participate will sign the ICF before undergoing any screening procedure. The screening period begins on the date the ICF is signed. Screening evaluations may be repeated as needed within the screening period; the investigator will assess patient eligibility according to the latest screening assessment results.

Results of standard-of-care tests or examinations performed before obtaining informed consent and  $\leq$  28 days before enrollment may be used for the purposes of screening rather than repeating the standard-of-care tests unless otherwise indicated. Voluntary, written informed consent for participation in the study must be obtained before any study-specific procedures are performed. ICFs for enrolled patients and for patients who are screened but not enrolled will be maintained at the study site.

All screening evaluations must be completed and reviewed to confirm that patients meet all eligibility criteria before enrollment. The investigator will maintain a screening log to record details of all patients screened and to confirm eligibility or record reasons for screening failure, as applicable.

During the Screening Visit, a complete physical examination will be conducted, including evaluations of: Head, eyes, ears, nose, and throat, Cardiovascular, Dermatological, Musculoskeletal, Respiratory, Gastrointestinal and Neurological systems

Any abnormality identified during screening will be graded according to NCI-CTCAE v5.0 and recorded. At subsequent visits (and as clinically indicated), limited, symptom-directed physical examinations will be performed. New or worsened clinically significant abnormalities are to be recorded as AEs.

The tissue biomarker sample collection schedule is described in Appendix 1 and in the Schedule of Assessments in each subprotocol (after screening).

Archival tumor tissues should consist of Formalin-Fixed Paraffin Embedded (FFPE) blocks or approximately 15 freshly cut unstained slides. If no archival tumor tissues are available, a fresh tumor biopsy at baseline (during screening period) is mandatory.

Blood samples will be taken predose on Day 1 to measure the circulating plasma EBV-DNA and other correlative markers as detailed.

## Table 1

| Assessment | Screening <sup>a</sup> | Notes |
|---|---|---|
| Days | -28 to ~ -1 | |
| Informed consent | х | |
| Inclusion/exclusion criteria | х | |
| Enrollment | x | |
| Demographics/medical history/prior medications | x | Includes age or year of birth, gender, self-reported race/ethnicity, tobacco consumption (ie, former or current or never) and history of treatment for the primary diagnosis, including prior medication, locoregional treatment plan. Information on radiographic studies performed before study entry may be collected for review by the investigator. Preexisting AEs at baseline should be recorded as medical history. |
| Vital signs/ height and weight | х | Vital signs include body temperature, pulse rate, and blood pressure (systolic and diastolic). Pulse rate and blood pressure will be collected. |
| Physical examination | х | A complete physical examination is required. |
| ECOG Performance<br>Status | х | |
| Adverse events | х | After the informed consent form has been signed but before the first administration of any study drug, only SAEs should be recorded. |
| Concomitant medications | х | |
| Hematology | X <sup>a</sup> | Local laboratory assessments on hematology, serum chemistry, coagulation parameters, and |
| Serum chemistry | Xª | urinalysis will be conducted, of which certain elements will be collected. |

| Assessment | Screening | Notes |
|---|---|---|
| Days | -28 to ~ -1 | |
| Fresh tumor tissue | x | Pre treatment Tissue will be collected either at time of diagnosis or after diagnosis, prior to to starting treatment. |

## 4.3.1 Screening Visits and Procedures

Patient accrual will be in accordance to the following chart showed in Figure 3. Only NPC patients whom have not previously received CRT treatment for NPC will be eligible for the clinical trial.

In addition, they must meet all inclusion criteria and do not fall within the exclusion criteria will be invited to give consent to participate in this clinical trial. After consent is given, the NPC patients will be accrued to start the trial.

## 4.3.2 Study Visits and Procedures

- 1. All patients undergoing the trial will undergo conventional CRT as the standard treatment for NPC.
- 2. For patients whom are accrued for the Phase 1 study, the dose of NK cells used in the treatment will be the same as the dose be evaluated in the determination of MTD. Once MTD is established, it will be used as the dose for all patients accrued subsequently.
- 3. Under the standard of care NPC treatment, chemotherapy will be carried out on week 1 and week 4. In addition, radiation treatment will be implemented daily Monday to Friday (2 Gyc per day) on week 1, 2, 3, 4, 5 and 6.
- 4. NK cells will be infused intravenously on week 3, 6, 7, 8, 9 and 10.
- 5. Interlukin-2 (200U/ml) will be co-administered with NK cells Plasma-Lyte148 supplemented with 2% HSA as a single infusion preparation.
- 6. A tumor tissue biopsy will be taken at screening period (<28 days before starting treatment) and at 11.
- 7. Blood (20 ml) will be taken at screening period (<28 days before starting treatment) before treatment starts (week 0) and at week 4, 7, 9 and 11.
- 8. For patients who are undergoing supplementary NK treatment at the end of the trial, four additional doses of NK cells will be infused by their early dosage respectively once a week on week 12, 13, 14 and 15.
- 9. For patients receiving supplementary NK cells treatment, an additional blood (20 ml) and tumor tissue biopsy will be taken on week 16.



Table 2

| Assessment<br>Period | Assessment Procedures | Notes |
|---|---|---|
| -28 to -1 | 1. Draw Blood (20ml) | |
| | 2. Tumor Tissue Biopsy | |
| | 3. EBV assay | |
| Week 1 | Chemo-drug Administration | |
| | <ol><li>Radiation Therapy Administration</li></ol> | |
| | (1 dose daily, 5 doses/week) | |
| Week 2 | <ol> <li>Radiation Therapy Administration</li> </ol> | |
| | (1 dose daily, 5 doses/week) | |
| Week 3 | Radiation Therapy Administration | |
| | (1 dose daily, 5 doses/week) | |
| | 2. NK cells infusion (NK cells + | |
| | Plasma-Lyte148 + IL-2 (200IU/ml) + | |
| | 2% HSA) | |
| Week 4 | 1. Draw Blood (20ml)* | *Draw blood before |
| | 2. EBV assay | Chemo-drug |
| | <ol><li>Chemo-drug Administration</li></ol> | administration but they |
| | <ol><li>Radiation Therapy Administration</li></ol> | may not be on the same |
| | (1 dose daily, 5 doses/week) | day. |
| Week 5 | Radiation Therapy Administration | |
| | (1 dose daily, 5 doses/week) | |
| Week 6 | Radiation Therapy Administration | |
| | (1 dose daily, 5 doses/week) | |

| | 2. NK cells infusion (NK cells + Plasma-Lyte148 + IL-2 (200IU/ml) + 2% HSA) | |
|---|---|---|
| Week 7 | <ol> <li>Draw Blood (20ml)*</li> <li>EBV assay</li> <li>NK cells infusion (NK cells + Plasma-Lyte148 + IL-2 (200IU/ml) + 2% HSA)</li> </ol> | *Draw blood before NK cells infusion but they ay not be on the same day. |
| Week 8 | 1. NK cells infusion (NK cells + Plasma-Lyte148 + IL-2 (200IU/ml) + 2% HSA) | |
| Week 9 | <ol> <li>Draw Blood (20ml)*</li> <li>EBV assay</li> <li>NK cells infusion (NK cell + Plasma-<br/>Lyte148 + IL-2 (200IU/ml) + 2%<br/>HSA)</li> </ol> | *Draw blood before NK cells infusion but they ay not be on the same day. |
| Week 10 | 1. NK cells infusion (NK cells + Plasma-Lyte148 + IL-2 (200IU/ml) + 2% HSA) | |
| Week 11 | <ol> <li>Draw Blood (20ml)</li> <li>Tumor Tissue Biopsy</li> <li>EBV assay</li> </ol> | |
| Week 12<br>(Optional) | NK cells infusion (NK cell + Plasma-<br>Lyte148 + IL-2 (200IU/ml) + 2%<br>HSA) | |
| Week 13<br>(Optional) | NK cells infusion (NK cell + Plasma-<br>Lyte148 + IL-2 (200IU/ml) + 2%<br>HSA) | |
| Week 14<br>(Optional) | NK cells infusion (NK cell + Plasma-<br>Lyte148 + IL-2 (200IU/ml) + 2%<br>HSA) | |
| Week 15<br>(Optional) | NK cells infusion (NK cell + Plasma-<br>Lyte148 + IL-2 (200IU/ml) + 2%<br>HSA) | |
| Week 16<br>(Optional) | <ol> <li>Draw Blood (20ml)</li> <li>Tumor Tissue Biopsy</li> <li>EBV assay</li> </ol> | |

## 4.3.3 Final Study Visit:

At the end of the trial, the patients will be reviewed for theirtolerability and safety of the allogeneic NK cell infusion.

## 4.3.4 Post Study Follow up and Procedures

As part of standard of care NPC surveillance protocol, both clinical and radiological assessments will be performed as follow:

- a) Clinical Assessments: Physical examination (including flexible nasopharyngoscopy to examine the nasopharynx) will be performed monthly for the first year and bi-monthly for the second and third year as part of the routine NPC surveillance protocol.
- b) Radiological Assessments: Baseline radiological imaging for tumor assessment and staging will be performed. Post-treatment radiological imaging will also be performed at 4-6 months post completion of treatment. Subsequent radiological studies will be performed as clinically indicated, determined by the treating physicians. The Response Evaluation Criteria in Solid Tumors (RECIST 1.1 criteria) will be used for assessment of response to therapy (from baseline to 4-6 month post treatment scans).

#### 4.4 Discontinuation/Withdrawal

#### 4.4.1 Discontinuation Criteria

Withdrawal Criteria:

- 1. Documented disease progression
- 2. Death
- 3. Development of an unacceptable toxicity, which in the opinion of the PIs, would render continued participation harmful.
- 4. Research subject or LAR withdraws consent from the study.
- 5. Investigator withdraws the subject from the study, in subject's best interest.
- 6. Non-compliance with protocol medications/administrations and/or required follow-up as judged by the PI.
- 7. Unable to be contacted and/or effectively monitored by the PIs and/or designees for follow-up (lost to follow-up).
- 8. Unable to receive the study infusion due to development of a significant health disorder, which in the judgment of the PI, would make proceeding with this study intervention to be not in the best medical interest of the participant.
- 9. Receipt of any therapy specifically for treatment of primary disease not defined in this protocol.

## 4.4.2 Discontinuation Visit and Procedures

Subjects may also withdraw voluntarily from receiving the study intervention for any reason during the study and they will continue to receive standard of care treatment for their cancer and follow up. Patients who withdraw from the study can give consent for their archival tissue samples to be used for correlative analyses with those who have completed the trial

#### 5 TRIAL MATERIALS

## 5.1 Trial Product (s)

#### 5.1.1. Cell Source

The source of the allogeneic NK cells are derived three sources:

- 1) Healthy Donor from the public
- 2) Donor from Patient's healthy relatives
- 3) GMP graded leukopaks.

The donor's eligibility criteria are as follows:

Gender: No preferenceAge: 21–50 years

Body Mass Index (BMI): 19.0–30.0 kg/m²

Haemoglobin level: 1) Female: > 12.5 g/dL; 2) Male: > 13g/dL

• Race/Ethnicity: No preference

Blood Group/Rh Type: No preference

• Pregnancy: Excluded

History of Malignancy: Excluded

## 5.1.2 Screening and Pre-Donation Requirements

Potential donors will be screened within seven days prior to the schedule donation date. Individuals who have undergone blood transfusion or major surgery or who have had any contagious disease in the past 6 months will be excluded. Donors must also refrain from taking any medications for at least 48 hours prior to blood collection.

## 5.1.3 Infectious Disease Testing

Each potential donor will be tested and confirmed negative for infectious disease within seven (7) days of donation:

- HIV-1/2 antigen and antibody
- Human T-lymphotropic virus types I/II (HTLV-I/II)
- Syphilis
- Cytomegalovirus (CMV) IgM and IgG
- Hepatitis B virus (HBV), Hepatitis C virus (HCV), and Hepatitis E virus (HEV)
- Vesicular stomatitis virus (VSV) IgG

#### 5.1.4. Collection and Handling

Approximately 300–400 mL of whole blood will be collected per donation using EDTA-containing infusion bags. All collected units will be transported immediately to the designated GMP facility for isolation of peripheral blood mononuclear cells (PBMCs). The isolated PBMCs will be aliquoted, freeze in CS10 media and store in Liquid Nitrogen. Approximately 300–400 mL of whole blood will be collected per donation using EDTA-containing infusion bags. All collected units will be transported immediately to the designated GMP facility for isolation of peripheral blood

mononuclear cells (PBMCs). The isolated PBMCs will be aliquoted, freeze in CS10 media and store in Liquid Nitrogen.

## 5.1.5. Allogeneic NK cells

Manufacturing of the Allogenic NK cells will be performed by ACTRIS- our national cell manufacturing facility.

This process includes:

- 1. Isolation of PBMC from whole blood
- 2. Enrichment and Expansion of NK cells from the isolated PBMCs
- 3. Preparation and formulation of Allogenic NK cells

## A. Work Flow of NK cell Manufacturing:

The NK cell Manufacturing workflow is shown in the flow diagram below.



- 1. Blood is obtained from consented healthy relative of cancer patients (300 ml 400ml); consented healthy public donor (300-400ml); and Commercial GMP leukopaks.
- 2. PBMC will be isolated from whole blood via SepMate 50.
- 3. The isolated PBMC will be analysed for 1) Sterility test.
- 4. For PBMC will be aliquot and freezed at 1x108 cells/ml per cryovial 5x106 cells/cryovial.
- 5. For batches of PBMC that did not clear the sterility test will be disposed in compliance with the Institutional guidance.
- 6. When sufficient PBMC cells are accumulated, they will be thawed and undergo NK cells enrichment using the Prodigy system.
- 7. The NK cells enrichment is achieved using CliniMACS CD3/CD56 complete kit used in conjunction with the Prodigy system.
- 8. After enrichment, A sample of the purified NK cells will undergo the Viability and Composition test.
- 9. The purified NK cells will be used for in-vitro NK cells expansion.
- 10. Expansion of NK cells will be carried out in G-Rex Bioreactors.

- 11. Cell count will be determined once a week.
- 12. After 14 dsays, NK cells will be harvested and seeded to multiple G-Rex Bioreactors to enable further growth.
- 13. 7-10 days later, NK cells will be harvested for QC testing.
- 14. Spent medium (40mL) will be sent for sterility test.
- 15. Also, samples of cells will tested sfor 1) Purity and 2) Viability as well as a 3) cell count.
- 16. Then, expanded NK cells will be aliquoted and freezed at 5x108 cells/ml in 20 mls of CS19 CS10 per freezing bag.
- 17. On the day of NK cells infusion, sufficient bags of cryo-preserved expanded NK cells will be thawed and diluted 10X volume of 0.9% saline supplemented with 5% Human serum albumin (HSA).
- 18. Centrifuge the thawed NK cells (500xg, 10 mins, 4oC) to pelletize the cells. Then, the supernatant is removed.
- 19. A small sample of the thawed NK cells will undergo test for 1) purity and 2) Viability.
- 20. Resuspend the rest of the NK cells into infusion media (Plasma-Lyte148, HSA (2%), IL-2(200IU/ml)).
- 21. Store the cells at 4oC (no more than 6 hours).
- 22. If the viability of the NK cells <70%, NK cells viability can be increased via counterflow centrifugation using the Rotea system.
- 23. Any excess expanded NK cells will be passed to the research lab.

## **B.** Manufacturing Methodologies

## i. Isolation of PBMC from whole blood:

#### Materials:

- The source of Blood will be from A) consented healthy relative of cancer patients (300 400 ml); B) Consented healthy public donor (300-400ml); C) Commercial GMP leukopaks.
- SepMate 50 (StemCell Technologies, cat no: 86450).
- Ficoll-Paque Premium density grandient medium (Cytiva, cat no: 17544202)
- CryoStor CS10 freezing medium (Biolife solutions, cat no: 210102)
- TheraPEAK PBS buffer (Lonza Bioscience, cat no: BEBP17-516Q)
- Human Serum Albumin (SK Plasma, cat no: 1D24E017SG)

#### Methods:

- 1) Add 15 ml of Ficoll-Paque into the SepMate<sup>™</sup> tube by carefully pipetting it through the central hole of the SepMate<sup>™</sup> insert. The top of the density gradient medium will be above the insert.
- 2) Dilute the whole blood with an equal volume of PBS + 2% human serum albumin and mix gently.
- 3) Keeping the SepMate<sup>™</sup> tube vertical, add the diluted whole blood by pipetting it down the side of the tube. The diluted whole blood will mix with the lymphoprep above the insert.
- 4) Centrifuge at 1200 x g for 10 minutes at room temperature, with the brake on.
- 5) Pour off the top layer, which contains the enriched PBMCs, into a new tube. Do not hold the SepMate<sup>™</sup> tube in the inverted position for longer than 2 seconds.
- 6) Wash the PBMC layer with 4 volume of 1xPBS supplemented with 2% human serum albumin.
- 7) Pelletize the PBMC (600xg, 10 min, RT).

- 8) Resuspend in NK MACS medium.
- 9) Draw a sample to perform a viable cell count followed by pelletization of the PBMC (600xg, 10 min, RT).
- 10) Remove the supernatant for sterility test.
- 11) Resuspend in CS10, aliquot and freeze the PBMC at 1x10<sup>8</sup> cells/ml per cryovial.

## ii. NK cells Enrichment and Expansion:

#### Materials:

- NK MACS GMP Medium (Mltenyi Biotec, catalog no. 170-076-356)
- CliniMACS CD3/CD56 complete kit (Miltenyi Biotec, cat no: 200-074-004)
- Human Serum Albumin (SK Plasma)
- IgG solution (SK Plasma)
- Sterile water for injection (B. Braun Medical Inc)
- GMP Human AB Serum (Akron Bio, catalog no: AR1010-0100)
- GMP IL-2 (Proleukin)
- Soluable MICA protein (SinoBiological, cat no: 12302-H08H)
- G-Rex 100M Bioreactor (WilsonWolf, cat no: 81100)
- Single use disposable Heamocytometer (Incyto, cat no: DHC-N01)
- Trypan blue solution, 0.4% (Bio-Rad, cat no. 1450021)
- CryoStor CS10 freezing medium (Biolife solutions, cat no: 210102)
- T175 culture flasks (Thermofisher Scientific, cat no: 159910)
- CryoMACS freezing bag 50 (Miltenyi Biotec, cat no: 200-074-400)
- Plasma-Lyte148 solution

#### Method:

| | Steps |
|---|---|
| Day 0 | <ol> <li>Frozen 20x10<sup>9</sup> PBMC cells are thawed.</li> <li>Change the cell suspension medium to NK MACS media without Serum and layer them on the treated surface to partially remove monocytes. 20 mls of the cell suspension is layer into each T175 flask with treated surface.</li> <li>Pooled the PBMC cells in NK MACS media.</li> <li>Introduce the suspended PBMC cells into the CliniMACS Prodigy system for automated NK cells enrichment using the CliniMACS CD3/CD56 complete kit.</li> <li>Collect a sample of total NK cells for Purity and Viability determination using Flow analysis.</li> <li>Also, the purified NK cells will undergo a viable cell count to ascertain the total number of NK cells.</li> <li>Then, 200x10<sup>6</sup> purified NK cells are pelletized by centrifugation (300xg, 5 min, RT) follow by resuspension in 200mL of NK Growth Medium supplemented wit Human AB Serum (5%), IL-2 (200 IU/ml) and soluble MICA (sMICA) (50ng/ml) to a final concentration of 1x10<sup>6</sup> NK cells/ml.</li> </ol> |

| | <ul> <li>8. The re-suspended NK cells are introduce into the G-Rex100M bioreactor before placing the bioreactor into an CO<sub>2</sub> incubator.</li> <li>9. The culture condition is to be maintained at 37°C, 5% CO<sub>2</sub>.</li> <li>10. Growing NK cells will settle at the bottom of the bioreactor to undergo proliferation.</li> </ul> |
|---|---|
| Day 3 | <ol> <li>Perform a viable NK cell count.</li> <li>Add 800mL of fresh NK MACS media supplemented with 5% human AB serum and 200IU/ml IL-2.</li> <li>After the addition, the total culture volume is 1000mL.</li> </ol> |
| Days 7 | <ol> <li>NK cell count will be performed once weekly.</li> <li>To perform a viable NK cell count, 800mL of the spent medium in the G-Rex100M Bioreactor are remove first.</li> <li>NK cells at the bottom will be mixed in the residual 200mL of medium.</li> <li>A sample is then taken for cell count.</li> <li>The cell number is estimated by trypan blue exclusion method with a heamocytometer.</li> <li>The 800mL removed in Step 2 will be put back into the G-Rex Bioreactor to enable further culture.</li> </ol> |
| Day 14 | <ol> <li>A viable NK cells cell count is performed as outlined at Day 7.</li> <li>If the NK number is above 200x10<sup>6</sup> cells, NK cell culture will divide into new G-Rex100M bioreactor by seeding the cells at 2 X 10<sup>6</sup> cells/cm<sup>2</sup> per bioreactor. All the G-Rex bioreactors will be top up with medium to 1000mL for further culture for another 7-10 days.</li> </ol> |
| Day 21 | <ol> <li>Perform a viable NK cell count as outlined at Day 7.</li> <li>If the NK cell number is still within exponential growth phase, the culture will be carried on for another 3 days.</li> <li>Otherwise, the NK cells will be harvested.</li> <li>During NK cells harvesting, 40mL of spend medium is collected for Sterility test.</li> <li>A cell sample is collected for purity and viability determination by flow cytometry.</li> <li>Another cell sample is collected for cytotoxicity assay to be performed in a non GMP laboratory.</li> <li>The rest of the NK cells will be labelled, aliquot and freeze in CS10 of 250 × 10<sup>6</sup> cells per 20 mL or 5 × 10<sup>7</sup> cells per bag for cryopreservation in each bag.</li> <li>The bags are cryopreserved and stored, ready to be use.</li> </ol> |

#### iii NK cells preparation for infusion:

# Day of infusion

- 1. Thawed sufficient cryo-preserved NK cells for infusion.
- 2. Dilute the thawed NK cells with 10x volume of Washing buffer (Saline solution, HSA(5%))
- 3. Centrifuge (500xg, 10min,4°C) to pelletize the NK cells.
- 4. Remove the supernatant containing DMSO.
- 5. Resuspend the NK cells in infusion media (Plasma-Lyte148, HSA(2%), IL-2(200IU/mI)).
- 6. Take a sample to analyze the purity and viability.
- 7. As a risk minimizing step, if the viability falls below the range of 40% 70%, the viability is increase through counterflow centrifugation via the Rotea system.
- 8. Keep the NK cells in infusion bag at 4°C (no more than 6 hr).

#### C. Sterility Test:

The cell culture Sterility assay will be out-sourced to TUV Ltd. In this assay, the cell culture media is to be determined for the absence of the following:

- Mycoplasma
- Endotoxin
- Sterility

## D. Purity and Viability Test:

The purity and viability of the expanded NK cells is determine by Flow Cytometry Analysis. In brief, approximately 1x10<sup>6</sup> NK cells from the expansion will be stained for CD56 (Miltenyi Biotec, cat no: 130-114-549), CD3 (Miltenyi Biotec, cat no: 130-114-710, and 7AAD Viability Dye (Miltenyi Biotec, cat no: 130-111-568). After staining, the purity and viability of NK cells can be calculated.

#### 5.2 STORAGE AND PRODUCT ACCOUNTABILITY

#### A. Storage:

- Allogeneic NK cells must be stored in a cryopreserved state at ≤ -150°C (e.g., vapor phase of liquid nitrogen) to maintain viability and functionality.
- Upon thawing, cells should be used immediately or within a specified short window (typically within **6 hours** at 2–8°C) to preserve cell quality.
- Avoid repeated freeze-thaw cycles to prevent loss of viability.

#### B. Label Elements on the Investigator Product

- Product Identification: AlloNK1 Allogenic NK cells
- Description: Allogenic expanded NK cells derived from healthy donor PBMCs
- Batch/Lot number: Unique identifier for traceability (each manufacturing run).:
- Study Protocol Number/Code: The clinical trial identifier
- Statement "For Investigational Use only"

- Route of Administration: For intravenous infusion only
- Storage Conditions: Store at 2–8 °C. Do not freeze and protect from light.
- Date of Manufacture / Expiration: Date of Manufacture, Date of Expiration
- Quantity/ Volume/ Cell Dose: Total cell number, total volume and the dosage
- Sponsor Name & Contact: Dr Lim Chwee Ming, (65) 98247996
- Subject identification number: Unique subject ID would be provided
- **Cohort number:** The cohort number the patient is enrolled into (eg: Phase 1 cohort 2)
- **Treatment number:** Treatment number indicates the sequence of dose a participant receives.
- Handling/ Special Precautions: Handle using aseptic technique and for allogenic use only
- **Disposal of NK cells:** Any unused, or nonconforming NK cell products will be disposed according to institutional and regulatory guidance. If the NK product is expired it would be returned back to the research lab of the study team.
- Instruction of Use: See Investigator's Brochure for administration instructions

#### C. Shipping:

- Cryopreserved NK cell products must be shipped in validated dry vapor shippers that maintain temperatures at or below -150°C throughout transit.
- Shipping containers must be equipped with temperature monitoring devices to document temperature stability during transport.
- Shipping must be coordinated to ensure timely delivery and immediate transfer to appropriate storage upon receipt.
- Shipping documentation must include product identification, batch number, storage instructions, and emergency contact information.

#### D. Disposal of Investigational Product on site

- Any unused, or nonconforming NK cell products must be disposed of following institutional and regulatory biosafety guidelines for biohazardous materials.
- Disposal procedures should ensure inactivation of viable cells through validated methods (e.g., autoclaving, chemical disinfection).
- All disposal activities must be documented, and records maintained in accordance with applicable regulations.

#### E. Disposal of Expired Investigational Product

 Any expired NK cell products will be transferred to our research lab to be used for preclinical investigation.

#### **6 TREATMENT**

#### 6.1 Rationale for Selection of Dose

In this trial, allogeneic NK cells are being used to add onto the standard chemoradiotherapy for NPC. The Maximum Tolerated Dose (MTD) will be between  $0.5 \times 10^7$  to  $1.8 \times 10^7$  NK cells/Kg (equivalent to approximately 0.5 to 1.0 billion NK cells). This dosage range of allogeneic NK cells is selected based on several Phase I cancer studies as a guide [7-10]. In these Phase I studies using allogeneic NK cells as the sole therapeutics, the dosage of allogeneic NK cells in the range of 1- 3 billions allogeneic NK cells exhibiting well tolerance. Therefore, in this Phase I trial with the infusion of allogeneic NK cells complementing standard chemoradiotherapy, we have proposed a

lower dose of  $0.5x10^7$  to  $1.8x10^7$  NK cells/Kg (equivalent to approximately 0.5 to 1.0 billion NK cells)

## **6.2 Study Drug Formulations**

The NK cells to be infused into NPC patients will undergo a media change to infusion media (Plasma-Lyte148, 2% human serum albumin, Interleukin-2 (200 Units/ml)) before transferred into in infusion bag and will be stored at 4°C (no more than 6 hr).

## 6.3 Study Drug Administration

Six doses of allogeneic NK cells at MTD will be administered for every accrued patient at during and after the radiotherapy via intravenous injection. Intravenous injection is selected because the intended target of the infused allogeneic NK cells is the small NPC cell clusters which are generated from the solid NPC tumor that are circulating in the blood during and after radiotherapy. The allogeneic NK cells infused into each patient will be derived from the PBMC of heatlhy volunteers.

## 6.4 Specific Restrictions / Requirements

In the event of an infusion related reaction, the patient may be treated accordingly although steroids should be avoided if possible (though not absolutely contraindicated). The use of agents such as H2 antagonists, antihistamines, acetaminophen, etc. is permitted for the treatment of infusion reactions. After appropriate treatment and resolution of the infusion reaction, NK cell infusion may be resumed at the discretion of the treating physician.

## 6.5 Monitoring Requirements

| Parameter | Timing/Frequency | Notes |
|---|---|---|
| Vital signs (temperature, blood pressure, heart rate, respiratory rate, oxygen saturation) | Before, during, and after<br>each NK cell infusion (e.g.,<br>baseline, 15 min, 30 min, 1<br>h, 2 h post-infusion) | Monitor for infusion<br>allergic reactions,<br>hypotension,<br>fever/chills. |
| Complete blood count (CBC) with differential & platelets | Baseline, then at least<br>twice weekly during<br>chemoradiotherapy, and<br>prior to each NK cell<br>infusion | Detect cytopenia<br>from CRT |
| Comprehensive<br>metabolic panel (liver<br>enzymes, renal function,<br>electrolytes) | Baseline, weekly or more frequently if abnormal | Monitor for hepatic/renal toxicity. |
| Coagulation profile (PT, aPTT, fibrinogen) | Baseline and as clinically indicated | Evaluate for coagulopathy and possible CRS or infection. |

| Infection screening<br>(blood cultures,<br>CRP/procalcitonin if<br>febrile) | Baseline and as clinically indicated | Example for rare rick of neutropenic infection. |
|---|---|---|
| Immune parameters (NK cell counts, cytokine panels, EBV DNA load) | Baseline, then specified time points post-infusion | Monitor NK persistence, immune activation, EBV viral load in NPC context. |
| Cardiac monitoring<br>(ECG, troponin,<br>echocardiogram | Baseline and if any symptoms | Recommended if<br>CRT includes<br>cardiotoxic agents<br>or for severe CRS |
| Neurological checks | Daily during<br>hospitalization; at each<br>visit outpatient | Watch for neurotoxicity (rare). |

## 6.6 Concomitant and adjuvant therapy

NK cells infusion will be administered concurrently (2 doses) and 4-6 doses as adjuvant dose.

## **7 SAFETY MEASUREMENTS**

## 7.1 Definitions

An adverse event (AE) is any untoward medical occurrence in a trial participant administered the NK cell product and may not necessarily have a causal relationship with this treatment.

An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the NK cell product.

A serious adverse event (SAE) is any untoward medical occurrence that at any dose:

- results in death
- is life-threatening
- requires inpatient hospitalisation or prolongation of existing hospitalisation
- results in persistent or significant disability/incapacity, or
- is a congenital anomaly/birth defect

## 7.2 Collecting, Recording and Reporting of Serious Adverse Events (SAEs) to CIRB

The reporting requirements will be in accordance to the reporting requirements published on CIRB website at the time when the event took place.

Only related SAEs (definitely/ probably/ possibly) will be reported to CIRB. Related means there is a reasonable possibility that the event may have been caused by participation in the clinical trial.

The investigator is responsible for informing CIRB after first knowledge that the case qualifies for reporting. Follow-up information will be actively sought and submitted as it becomes available.

Related AEs will not be reported to CIRB. However, the investigator is responsible to keep record of such AEs cases at the Study Site File.

# 7.3 Collecting, Recording and Reporting of Serious Adverse Events (SAEs) to the Health Sciences Authority (HSA)

The investigator will assess the severity of each AE and SAE reported during the study. AEs and SAEs should be assessed and graded based upon NCI-CTCAE v5.0.

Toxicities that are not specified in NCI-CTCAE will be defined as follows:

- Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated
- Grade 2: Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL)
- Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL
- Grade 4: Life-threatening consequences; urgent intervention indicated
- Grade 5: Death related to AE

#### The following are **not** considered to be SAEs:

- Hospitalization for elective treatment of a preexisting condition that did not worsen from baseline
- Hospitalization for social/convenience considerations
- Scheduled therapy for the target disease of the study, including admissions for transfusion support or convenience

The assessment of study drug relationship to each AE will be reported on the appropriate source document (and SAE form, in the event of an SAE) by the Investigator or designee according to his or her best clinical judgment. The criteria listed in Table 3 should be used to guide this assessment. Please note that not all criteria must be present to be indicative of a particular drug relationship.

In this study, imAEs are of special interest. Potential imAEs are listed in Table 3 below.

**Table 3: Adverse Event Causality Guidelines** 

| Body System Affected | Events |
|----------------------|--------|
|----------------------|--------|

| Skin (mild-common) | pruritus or maculopapular rash; vitiligo |
|---|---|
| Skin (moderate) | follicular or urticarial dermatitis; erythematous/lichenoid rash; Sweet syndrome |
| Skin (severe-rare) | full-thickness necrolysis/Stevens-Johnson syndrome |
| Gastrointestinal | colitis (includes diarrhoea with abdominal pain or endoscopic/radiographic evidence of inflammation); pancreatitis; hepatitis; ALT/AST elevation; bowel perforation |
| Endocrine | thyroiditis, hypothyroidism, hyperthyroidism; hypophysitis with features of hypopituitarism, eg, fatigue, weakness, weight gain; insulindependent diabetes mellitus; diabetic ketoacidosis; adrenal insufficiency |
| Respiratory | pneumonitis/diffuse alveolitis |
| Eye | episcleritis; conjunctivitis; iritis/uveitis |
| Musculoskeletal | arthritis; arthralgia; myalgia; myasthenic syndrome/myasthenia gravis; myositis |
| Blood | anemia; leukopenia; thrombocytopenia |
| Renal | interstitial nephritis; glomerulonephritis; acute renal failure |
| Cardiac | pericarditis; myocarditis; heart failure |
| Neurologic | encephalitis; Guillain-Barre syndrome; meningitis; meningoradiculitis; meningoencephalitis; neuropathy |

| Classification Definition |
|---------------------------|
|---------------------------|

| Likely Related | There is a clear temporal association between the event and the administration of study drug, a plausible mechanism for the event to be related to the study drug and causes other than the study drug has been ruled out, and/or the event re-appeared on re-exposure to the study drug. |
|---|---|
| Probably Related | The event is a known or suspected effect of the study drug and follows a reasonable temporal sequence from the administration of study drug but cannot be readily explained by study participant or study factors, and/or the event ceases or diminishes with discontinuation of study medication |
| Possibly Related | There is an association between the event and the administration of the study drug and there is a plausible mechanism for the event to be related to study drug, but there may also be alternative etiology, such as characteristics of the patient's clinical status or underlying disease. |
| Unlikely Related | The event is unlikely/remotely possible /probably not related to the study drug and likely to be related to factors other than the study drug. |
| Not Related | The event is related to an etiology other than the study drug (the alternative etiology must be documented in the study patient's medical record). |

## 7.4 Known or potential adverse event related to post-infusion of IP (AlloNK1)

Events that are undesirable but usually manageable or mild/moderate, without causing life-threatening risk, hospitalization, or permanent impairment such as the following:

- Infusion-related reactions (<5%): fever, chills, rigors, headache, mild hypotension.
- Mild Infections (<5%): uncomplicated bacterial/viral infection related to transient immunosuppression.
- Cytopenia (5-10%): neutropenia, anaemia, thrombocytopenia (usually CRT-related).
- Mild Hepatic/renal toxicities (<5%): Transient enzyme elevations or creatinine rise.</li>
- Mild Neurotoxicity (<1%): mild confusion without major sequelae.

## 7.5 Known or potential serious adverse event related to post-infusion of IP (AlloNK1)

Events that result in death, are life-threatening, require/prolong hospitalization, cause persistent disability, or are medically significant such as the following:

- Cytokine Release Syndrome (CRS): even if rare and milder than CAR-T cells, if it causes hypotension requiring vasopressors, high-grade fever, or ICU-level care, it will be considered as an SAE.
- Severe infections: presence of sepsis, pneumonia, or other infections requiring IV antibiotics or hospitalization.
- Graft-versus-host disease (GVHD): any clinically significant GVHD is considered an SAE.
- Hepatic/renal toxicities acute liver failure, grade 3–4 enzyme elevations, renal failure requiring dialysis.
- Neurotoxicity: seizures, encephalopathy, or any neurological event requiring intervention or hospitalization.
- Tumor lysis syndrome: especially if it leads to renal impairment, arrhythmia, or hospitalization.

## 7.6 Management of AE and SAE

Our team comprises of haematologists specializing in managing these cell therapy related complications indicated table 4:

Table 4

| Events | Recommended Management |
|---|---|
| Infusion reaction (mild–<br>moderate) | Pause/slow infusion, give antipyretics, antihistamines; monitor vitals closely. |
| CRS (grade ≥2) | Supportive care (IV fluids, oxygen), consider tocilizumab / corticosteroids as deemed appropriate by our haematologist. Escalate to HD or ICU care if hypotensive requiring vasopressors. |
| Infection | Prompt cultures, broad-spectrum antibiotics; prophylactic antimicrobials per institutional guidelines during neutropenia. |
| Cytopenia | Growth factor support (G-CSF), transfusions as indicated. |
| GVHD (if suspected) | Standard immunosuppressive therapy (high-dose steroids) and consult transplant/immune specialists. |
| Neurotoxicity | Supportive management, consider corticosteroids, seizure prophylaxis if indicated. |
| Tumor lysis / electrolyte abnormalities | Hydration, monitor electrolytes, rasburicase/allopurinol as per protocol. |

## 7.7 Safety Monitoring Plan

The principal investigator will be responsible for the safety and well-being of subjects, and integrity of data collected.

#### **Data and Safety Monitoring**

A safety review committee (SRC) will monitor the safety data during Phase 1 of the study on a periodic basis to help ensure the ongoing safety of study patients. The SRC will consist of at least 3 investigators of the study, a pharmacist and biostatistician. The SRC will meet regularly during the Phase 1 dose escalation portion of the study to review all accumulated available data, including safety and preliminary efficacy to make recommendations on continuation, modification, or suspension of the study. The SRC will make recommendations concerning dose escalation/deescalation or any changes to the dosing paradigm based on review of available data prior to proceeding to the next dose level. The SRC will also make recommendations about the dose selected for Phase 2 and overall study conduct.

## 7.8 Complaint Handling

Any compliant will be submitted to the SRC for their review process. A response will be provided within 21 days.

## **8 DATA ANALYSIS**

## 8.1Data Quality Assurance

Data will be collected and recorded by a clinical research coordinator. The investigator will verify that all data entries are accurate and correct, including verification that the subject fulfils the criteria for entry into the study before study treatment commences.

#### 8.2 Data Entry and Storage

All data obtained in the study described in this protocol will be recorded on paper case report forms (CRFs). The CRF for each subject will be presented in a folder. The CRF will be completed chronologically and updated regularly in order to reflect the most recent data on the patient included in the study.

Each CRF must be neatly filled in with a black-inked pen. For each page on which information is entered, the subject number must be recorded. CRFs will be dated and signed by an investigator.

Errors must be corrected by drawing a single line through the incorrect entry and by writing the new value as close as possible to the original. The correction must then be initialed and dated by an authorized study team member.

CRFs and Investigator Site Folder will be kept in a secure cabinet, under lock and key. Only members of the study team can have access to the data.

#### 9 SAMPLE SIZE AND STATISTICAL METHODS

#### 9.1 Determination of Sample Size

In the Phase I study, we will be using the Bayesian Model Averaging continual reassessment method (BMA-CRM) study design [12, 13]. The primary goal of the BMA-CRM is to identify the maximum tolerated dose (MTD) of NK cells to be infused. In this Phase I study, minimum of 21 patients will be accrued. Five doses of NK cells will be used (0.5x10<sup>7</sup>, 0.8x10<sup>7</sup>, 1.1x10<sup>7</sup>, 1.4x10<sup>7</sup> and 1.8x 10<sup>7</sup>cells/Kg). We will begin with the dose 0.8x10<sup>7</sup>cells/kg and the dose escalation is restricted to a single dose level. Once there is an occurrence of 1 toxicity, the CRM will be implemented. The CRM method estimates toxicity at each dose using Bayesian methodology to update a dose-toxicity curve for each cohort of 3 patients. We assume the prior toxicity probability estimates at 10%, 15%, 20%, and 25% at each level. To avoid subjectivity in setting priors, the BMA-CRM specifies multiple sets of priors and takes the average across the CRM models to avoid the potential estimation bias caused by misspecification. We shall terminate the phase at 21 patients or when CRM dictate that 6 patients be treated at a particular dose, at which point the current dose estimate is declared the MTD.

Phase 2 is a single-arm trial; the one-sample proportion test will be used to test the proportion deduction based on the binomial distribution. A sample size of 5 achieves 80.549% power to detect a difference (P1-P0) of -0.2500 using a one-sided exact test with a significance level (alpha) of 0.05. These results assume that the population proportion under the null hypothesis (P0) is 1.00. Assume the withdrawal rate at 0.2 (20%), the total sample size is estimated at 6. From phase 1a, for those patients treated at MTD, these patients will be followed up and included in the phase 2 study. As likely there will be around six patients treated at MTD (at least two cohorts), thus only an additional one patient will be included for the phase 2 trial.

## 9.2 Statistical and Analytical Plans

#### A. General Considerations:

The phase 1 study will be an open-label, dose-escalation trial, with a maximum of 21 NPC patients to be accrued for NK cells treatment. The primary endpoint is the occurrence of any of the toxicities during 4 weeks of treatment as assessed by AEs attributed (see session 7.3). Five doses of NK cells will be used for the treatment ( $d_1 = 0.5 \times 10^7$ ,  $d_2 = 0.8 \times 10^7$ ,  $d_3 = 1.1 \times 10^7$ ,  $d_4 = 1.4 \times 10^7$ , and  $d_5 = 1.8 \times 10^7$  cells/kg). The maximum tolerated dose (MTD) will be estimated as the highest dose with an estimated probability of a dose limiting toxicity (DLT) of less than 30%.

We will apply 2-stage continual reassessment method (CRM) design (Cheung 2005 & 2011; Goodman 1995). First, we specify a stage 1 design as a predetermined nondecreasing dose sequences. Because the 3+3 algorithm is familiar, we consider the "group-of-three" stage 1 design whereas escalation takes place after every group of three nontoxic outcomes. The stage 1 design is in effect until the first observed toxicity. Secondly, the trial turns to the model-based CRM for dose assignment. CRM method generally has a superior operating performance as it bases estimation on all prior dose data rather than just the last 3 patients; this usually resulted in more accurate estimation of the MTD, fewer toxicities and more patients treated at assumed efficacious doses close to the MTD.

#### Specifically, for stage 1:

The first three patients  $(x_{i,0})$  will be recruited at dose level  $d_2$ . Starting at  $d_2$  is because that NK cell treatments are given at established doses which is thought to be non-toxic.

If no DLT occurs, subsequent three patients will be recruited at one dose higher (unless current dose is D6).

$$x_{1,0} = x_{2,0} = x_{3,0} = d_2, x_{4,0} = x_{5,0} = x_{6,0} = d_3, \dots$$

The MTD will be estimated as the last dose ( $d_5$ ).

If a DLT occurs, the trial will progress to stage 2 using a CRM to assign the dose (see below).

#### For stage 2:

The study will progress to this stage if a DLT occurs in stage 1. We will assign 3 patients at a time to each does, and update the model-based estimates between every group of 3 patients, using information of all patients with DLTs known by the next patient recruitment time. Escalation by more than 1 level will not be allowed. If the number of consecutive patients on the current dose is 6 or 21 patients in total then the trial will stop and the MTD will be estimated based on a CRM of the recruited patients.

We use maximum likelihood estimation in conjunction with the CRM. The idea is analogous to the Bayesian CRM, with the data observed in the first i –1 patients. The dose for the next subject is computed based on the maximum likelihood estimates of coefficients for given data.

A CRM will be implemented via the function implemented in R package "dfcrm" [15]. The prior toxicity estimates are set at 2.5%, 5%, 10%, 20%, 30% for the dose levels from D1 to D6. We shall terminate the phase at 21 patients or when a dose level is selected 6 times at which point the current dose estimate is declared the MTD.

The properties of the CRM procedure are assessed using the CMR Suite v1.00 using simulated data [12, 13]. We assume patients recruited randomly, with average arrival of 1.25 per month, toxicity assessment period is within 30 days, and target toxicity limit (TTL) probability is 30%. The simulation is applied to 5 scenarios from true low to very high toxicity rates using 1000 replicates for each scenario. The table below compares the performance in each circumstance in terms of the total and an average number of DLT, the proportion of times each dose level is selected as MTD, the proportion of total patients treated at each dose level, and the duration of trial time. If the true toxicity is low, around 19.8 months are expected to complete the trial, and the toxicity per trial is low at 2.7, and MTD is estimated at the dose level 5.

#### Model

| Target Toxicity Probability | 0.300 |
|---------------------------------------------------------------------|-------|
| Safety Stopping Probability<br>(Upper Limit Pr(tox) at Lowest Dose) | 0.700 |
| Maximum Sample Size | 21 |
| Cohort Size | 3 |
| Starting Dose Level | 2 |

| Toxicity Assessment Period (Days) | 30 |
|-----------------------------------|----|
|-----------------------------------|----|

## Prior **Median** Probabilities of Toxicity at Each Dose Level:

| Dose | Prob. |
|------|-------|
| 1 | 0.025 |
| 2 | 0.050 |
| 3 | 0.100 |
| 4 | 0.200 |
| 5 | 0.300 |

## Scenarios and Results

## **Scenario: Very High Toxicity**

| Dose<br>Level | True Prob(tox) | Selection Probability | # of Subjects Treated | # of Toxicities |
|---|---|---|---|---|
| 1 | 0.200 | 0.11 | 1.7 | 0.4 |
| 2 | 0.300 | 0.24 | 7.3 | 2.2 |
| 3 | 0.400 | 0.22 | 4.6 | 1.8 |
| 4 | 0.500 | 0.07 | 1.5 | 0.7 |
| 5 | 0.600 | 0.01 | 0.2 | 0.1 |

**Probability of Early Termination:** 0.35

**Toxicities per Trial:** 5.2

Total Trial Time (Months): 15.65

## **Scenario: High Toxicity**

| Dose<br>Level | True Prob(tox) | Selection Probability | # of Subjects Treated | # of Toxicities |
|---|---|---|---|---|
| 1 | 0.100 | 0.03 | 0.8 | 0.1 |

| 2 | 0.200 | 0.17 | 6.7 | 1.4 |
|---|-------|------|-----|-----|
| 3 | 0.300 | 0.35 | 6.5 | 1.9 |
| 4 | 0.400 | 0.25 | 3.6 | 1.4 |
| 5 | 0.500 | 0.05 | 0.8 | 0.4 |

**Probability of Early Termination: 0.16** 

**Toxicities per Trial:** 5.2

Total Trial Time (Months): 19.01

## **Scenario: Medium Toxicity**

| Dose Level | True Prob(tox) | Selection Probability | # of Subjects Treated | # of Toxicities |
|---|---|---|---|---|
| 1 | 0.050 | 0.00 | 0.1 | 0.0 |
| 2 | 0.100 | 0.03 | 4.6 | 0.5 |
| 4 | 0.250 | 0.32 | 5.2 | 1.3 |
| 5 | 0.300 | 0.41 | 4.2 | 1.3 |

**Probability of Early Termination:** 0.04

**Toxicities per Trial:** 4.2

**Total Trial Time (Months): 20.55** 

## **Scenario: Low Toxicity**

| Dose<br>Level | True Prob(tox) | Selection Probability | # of Subjects Treated | # of Toxicities |
|---|---|---|---|---|
| 1 | 0.000 | 0.00 | 0.0 | 0.0 |
| 2 | 0.025 | 0.00 | 3.2 | 0.1 |
| 3 | 0.050 | 0.00 | 3.5 | 0.2 |
| 4 | 0.100 | 0.06 | 4.3 | 0.4 |
| 5 | 0.200 | 0.93 | 9.9 | 2.0 |

Probability of Early Termination: 0.01

Toxicities per Trial: 2.7

Total Trial Time (Months): 19.85

#### Phase 2:

#### Statistical Analysis and Power calculation (new to 10%)

The reference we use in comparison with our single arm trial finding is derived from the anticipated proportion of locally advanced NPC patients (25-30%) who will continue to present with detectable circulating EBV-DNA following standard of care CRT paradigm. We hypothesize that in this single arm trial, adding allogeneic NK cells will completely eliminate the proportion of patients with detectable circulating EBV-DNA from 25-30% to 10%. Hence, applying the one proportion Z-score test, a sample size of 26 will achieve 81.2% power to detect a difference (P1-P0) of 20% using a one-sided exact test with a significance level (alpha) of 0.05. Assuming the withdrawal rate at 0.2 (20%), the total sample size is estimated at 31. In our phase 1 design, at least 6 patients will be treated at our MTD of allogenic NK cells, meaning that additional 25 patients will be accrued in the phase 2 trial.

The proportion estimate and its confidence interval will also be reported. We will also perform sensitivity analyses to assess the impact of missing data and potential confounding variables.

The secondary endpoint of the study is to determine the change in patient survival and recurrence rate within 24-36 months post-treatment when compared with historic cohorts under standard treatments. This is an exploratory aim due to small sample size. We will apply Kaplan-Meier curves to plot the survival and recurrence rate with time. We will estimate the median and mean survival time, and the confidence intervals. The median survival time will be estimated. We will compare the survival and recurrence rates between the study cohort and the historical control group using log-rank tests.

#### **B. Safety Analyses**

The phase 1 study is safety-oriented design. Adverse events will be monitored and recorded throughout the study. Dose toxicity evaluation after receiving the treatment will be conducted. Dose escalation will occur only if no toxicity occurred or as suggested by CRM. Dose-limiting toxicities will be defined and recorded. We will also examine the proportion of patients who experience treatment-related adverse events and report them separately.

## 9.3 Interim Analyses

- The dose-escalation design CRM foresees that decisions based on the current data are taken before the end of the study. More precisely, after each cohort in the dose-escalation part, the next dose will be chosen depending on the observed data. The study may be stopped early if predefined stopping rules are met.
- At the mid-point of Phase 2, we will access the progress of our primary endpont by the determination of the percentage of patients achieving undectable EBV-DNA levels and secondary endpoint of recurrent rate among all the accrual for the trial thus far.

## 9.4 Describe the types of statistical interim analyses, including their timing

- See the analysis method session for CRM methods.
- A statistical two tailed test will be perform to examine the decrease in the percentage of patients with undectable EBV-DNA levels,
- Similar statistical analysis will be carried out to analyse the NPC recurrence rate among the accurals for the trial at the point of analysis.

#### 10 DIRECT ACCESS TO SOURCE DATA/DOCUMENTS

The investigator(s)/institution(s) will permit study-related monitoring, audits and/or IRB review and regulatory inspection(s), providing direct access to source data/document.

In accordance with ICH GCP guidelines, the study monitor must have direct access to the investigator's source documentation in order to verify the data recorded in the investigator file for consistency. The monitor is responsible for routine review of the investigator file at regular intervals throughout the study to verify adherence to the protocol and the completeness, consistency, and accuracy of the data being entered on them. The investigator agrees to cooperate with the monitor to ensure that any problems detected during these monitoring visits are resolved.

#### 11 QUALITY CONTROL AND QUALITY ASSURANCE

Data will be collected and recorded by a clinical research coordinator. The investigator will verify that all data entries are accurate and correct, including verification that the subject fulfils the criteria for entry into the study before study treatment commences.

#### 12 ETHICAL CONSIDERATIONS

This study will be conducted in accordance with the ethical principles that have their origin in the Declaration of Helsinki and that are consistent with the Good Clinical Practice and the applicable regulatory requirements.

This final Clinical Trial Protocol, including the final version of the Participant Information Sheet and Consent Form, must be approved in writing by the Centralised Institutional Review Board (CIRB) and regulatory approval from Health Sciences Authority (HSA), prior to enrolment of any patient into the study.

The principle investigator is responsible for informing the CIRB and HSA of any amendments to the protocol or other study-related documents, as per local requirement.

#### 12.1 Informed Consent

The study will be conducted in accordance with the protocol, International Conference on Harmonization (ICH) GCP guidelines, applicable regulations and guidelines governing clinical study conduct and ethical principles that have their origin in the Declaration of Helsinki. The investigator will ensure that the study is conducted in accordance with the provisions as stated in the ICH regulations and complies with prevailing local laws and customs. Prior to the initiation of any screening or study-specific procedures, the investigator and/or his/her representative will explain the nature of the study to the subject and answer all questions regarding this study. Each informed consent will be reviewed, signed and dated by the subject and the person who administered the informed consent. A copy of each informed consent will be given to the subject and each original will be placed in the Investigator Site Manual.

## 12.2 Confidentiality of Data and Patient Records

Information collected for this study will be kept confidential. This confidentiality is extended to cover testing of any biological samples and genetic tests in addition to the clinical information relating to the participating subjects. Patient records, to the extent of the applicable laws and regulations, will not be made publicly available. Data collected and entered into the Case Report Forms are the property of SGH. In the event of any publication regarding this study, patient identity will remain confidential.

#### 13 PUBLICATIONS

The investigators have the right to publish the results of the study, but with due regard to the protection of confidential information.

#### 14 RETENTION OF TRIAL DOCUMENTS

Records for all participants, including CRFs, all source documentation (containing evidence to study eligibility, history and physical findings, laboratory data, results of consultations, etc) as well as DSRB records and other regulatory documentation will be retained by the PI in a secure storage facility for up to 10 years from time of study termination. The records will be accessible for inspection and copying by authorized authorities.

#### 15 FUNDING AND INSURANCE

The Insurance is covered under the Singhealth Insurance policy for clinical trial in its terms and provisions, its legal liability for injuries caused to participating persons and arising out of this research performed strictly in accordance with the scientific protocol as well as with applicable law and professional standards. Since this is a first in man clinica trial, additional insurance will be acquired.

The funding is supported under the PI's National Medical Research Council. Clinician Scientist Award (CSA) and Clinical Trial Grant – Investigator Initiated trial (CTG-IIT).

## LIST OF ATTACHMENTS

## **Appendix 1 Study Schedule**



| Assessment<br>Period | Assessment Procedures | Notes |
|---|---|---|
| -28 to -1 | 1. Draw Blood (20ml) | |
| | Tumor Tissue Biopsy | |
| | 3. EBV assay | |
| Week 1 | <ol> <li>Chemo-drug Administration</li> <li>Radiation Therapy Administration<br/>(1 dose daily, 5 doses/week)</li> </ol> | |
| Week 2 | Radiation Therapy Administration (1 dose daily, 5 doses/week) | |
| Week 3 | <ol> <li>Radiation Therapy Administration (1 dose daily, 5 doses/week)</li> <li>NK cells infusion</li> </ol> | |
| Week 4 | <ol> <li>Draw Blood (20ml)*</li> <li>EBV assay</li> <li>Chemo-drug Administration</li> <li>Radiation Therapy Administration<br/>(1 dose daily, 5 doses/week)</li> </ol> | *Draw blood before<br>Chemo-drug<br>administration |
| Week 5 | Radiation Therapy Administration (1 dose daily, 5 doses/week) | |
| Week 6 | <ol> <li>Radiation Therapy Administration</li> <li>(1 dose daily, 5 doses/week)</li> <li>NK cells infusion</li> </ol> | |

| Week 7 | 1. Draw Blood (20ml)* 2. EBV assay 3. NK cells infusion | *Draw blood before NK cells infusion |
|---|---|---|
| Week 8 | NK cells infusion | |
| Week 9 | NK cells infusion | |
| Week 10 | NK cells infusion | |
| Week 11 | Draw Blood (20ml) Tumor Tissue Biopsy BV assay | |
| Week 12<br>(Optional) | NK cells infusion | |
| Week 13<br>(Optional) | NK cells infusion | |
| Week 14<br>(Optional) | NK cells infusion | |
| Week 15<br>(Optional) | NK cells infusion | |
| Week 16<br>(Optional) | <ol> <li>Draw Blood (20ml)</li> <li>Tumor Tissue Biopsy</li> <li>EBV assay</li> </ol> | |

## **NK cell infusion**

- 1. 6 doses will be administered during the standard of care treatment of concurrent chemoradiotherapy (2 doses as concurrent and 4 doses as adjuvant therapy).
- 2. The first 3 patients admitted for the administration of the first dose of NK cells will be monitored overnight. The expected duration of NK cell infusion is approximately 30-60 mins over a slow infusion. If there are no acute reactions to NK cell infusion for the first 3 patients, subsequent doses to the 3 patients can be treated as outpatient with a monitoring of 4-6 hours following infusion.
- 3. Without acute reaction, NK cells infusion for the rest of the patients accrued will be treated as outpatient with a monitoring of 4-6 hours following infusion
- Patients who have persistently detectable circulating plasma EBV-DNA copies after the 6
  doses of NK cell infusions will have the option of receiving an additional 4 weekly cycles
  of NK cells infusion.

#### **Radiation Therapy**

Conventional radiotherapy will be given as per standard of care treatment of NPC

## **Chemotherapy**

- 1. Platinum based chemotherapy regime is usually administered as the standard of care chemotherapy option for NPC.
- 2. In patients who cannot receive chemotherapy or declined chemotherapy option, they will still be eligible to participate in this trial.
- 3. Patients who are prescribed other chemotherapy beside the platinum based chemotherapy option due to adverse response to platinum chemotherapy are also eligible to participate in this trial.

## **Correlative tissue Biopsy and blood analyses**

- 1. A total of 2 tumor biopsies will be performed in this trial (once prior to treatment and the other after the completion of the standard treatment and 6 doses of NK cells infusion).
- 2. Blood (approximately 20 ml) will be drawn 5 times (prior to treatment, week 4, 7, 9 and 11) during the trial. Sufficient plasma will be send for plasma EBV detection and the rest will be frozen for analysis at a later stage.
- 3. PBMC will be isolated and stored for correlative analyses.

## References

- 1. Del Zotto, G., et al., *Markers and function of human NK cells in normal and pathological conditions*. Cytometry B Clin Cytom, 2017. **92**(2): p. 100-114.
- 2. Wu, J. and L.L. Lanier, *Natural killer cells and cancer*. Adv Cancer Res, 2003. **90**: p. 127-56.
- 3. Dianat-Moghadam, H., et al., *NK cells-directed therapies target circulating tumor cells and metastasis*. Cancer Lett, 2021. **497**: p. 41-53.
- 4. Han, B., et al., Altered NKp30, NKp46, NKG2D, and DNAM-1 Expression on Circulating NK Cells Is Associated with Tumor Progression in Human Gastric Cancer. J Immunol Res, 2018. **2018**: p. 6248590.
- 5. Myers, J.A. and J.S. Miller, *Exploring the NK cell platform for cancer immunotherapy*. Nat Rev Clin Oncol, 2021. **18**(2): p. 85-100.
- 6. Shimasaki, N., A. Jain, and D. Campana, *NK cells for cancer immunotherapy.* Nat Rev Drug Discov, 2020. **19**(3): p. 200-218.
- 7. Ciurea, S.O., et al., *Phase 1 clinical trial using mblL21 ex vivo-expanded donor-derived NK cells after haploidentical transplantation.* Blood, 2017. **130**(16): p. 1857-1868.
- 8. Hoogstad-van Evert, J., et al., Intraperitoneal infusion of ex vivo-cultured allogeneic NK cells in recurrent ovarian carcinoma patients (a phase I study). Medicine (Baltimore), 2019. **98**(5): p. e14290.
- 9. Ishikawa, T., et al., *Phase I clinical trial of adoptive transfer of expanded natural killer cells in combination with IgG1 antibody in patients with gastric or colorectal cancer.* Int J Cancer, 2018. **142**(12): p. 2599-2609.
- 10. Lin, M., et al., *Pembrolizumab plus allogeneic NK cells in advanced non-small cell lung cancer patients.* J Clin Invest, 2020. **130**(5): p. 2560-2569.
- 11. Jin, Y.Y., et al., Chemoradiotherapy combined with NK cell transfer in a patient with recurrent and metastatic nasopharyngeal carcinoma inducing long-term tumor control: A case report. Medicine (Baltimore), 2020. **99**(43): p. e22785.
- 12. O'Quigley, J., M. Pepe, and L. Fisher, *Continual reassessment method: a practical design for phase 1 clinical trials in cancer.* Biometrics, 1990. **46**(1): p. 33-48.
- 13. Yin, G. and Y. Yuan, *Bayesian model averaging continual reassessment method in phase I clinical trials*. Journal of the American Statistical Association, 2009. **104**(487): p. 954-968.
- 14. cheung, Y.K., *Coherence principles in dose-finding studies.* Biometrika, 2005. **92**: p. 10.
- 15. Cheung, Y.K., *Dose Flnding by the Continual Reassessment Method*. 2011: Chapman & Hall/CRC press.

| 16. | Goodman, S.N., M.L. Zahurak, and S. Piantadosi, <i>Some practical improvements in the continual reassessment method for phase I studies</i> . Stat Med, 1995. <b>14</b> (11): p. 1149-61. |
|---|---|